CLINICAL TRIAL: NCT05109013
Title: Juvenile Essential Arterial Hypertension and Vascular Reactivity in Systemic and Cerebral Circulation
Brief Title: Juvenile Essential Arterial Hypertension and Vascular Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Head of Department of Physiology and Immunology Faculty of Medicine Osijek, Josip Juraj Strossmayer University of Osijek
Other Study IDs: 2158-61-07-21-06
Record Dates: First submitted 2021-09-02; First posted 2021-11-05 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Child, Only; Essential Hypertension
Keywords: cerebral circulation; child; endothelium; microcirculation; macrocirculation; hypertension; oxidative stress
MeSH Terms: conditions — Essential Hypertension; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NT group - normotensive children
- HT group - hypertensive children

SUMMARY:
The main goal of this study is to investigate the association of the juvenile essential arterial hypertension with systemic micro- and macrovascular reactivity and cerebral vascular function, and to examine the potential impact of elevated oxidative stress on this associations.

ELIGIBILITY:
Inclusion Criteria:

* healthy normotensive children and children with essential arterial hypertension

Exclusion Criteria:

* secondary arterial hypertension
* other systemic diseases with immunopathology
* neurodegenerative diseasesat
* children that use therapy which has a high impact on vascular or immunological function (immunotherapy, immunosuppressive therapy, sistemic corticosteroid therapy etc..).

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children aged 9-18 years of both sexes; normotensive and children with essential arterial hypertension
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Systemic microvascular function in children | Day 1.
  Skin microvascular reactivity assessed by Laser Doppler flowmetry (post-occlusive reactive hyperemia, iontophoresis of acetylcholine and sodium nitroprusside) - measured in perfusion units (PU)
Systemic macrovascular function in children | Day 1.
  Vascular ultrasound measurement of brachial artery response to vascular occlusion (flow mediated dilation; FMD, %)
Cerabral vascular function in children | Day 1.
  Cerebral blood flow velocities assessed by transcranial Doppler sonography (cm/s)

SECONDARY OUTCOMES:
Oxidative stress - thiobarbituric acid reactive substances (TBARS) | Day 1.
  Serum sample collection for measurement of biomarkers of oxidative stress level. Thiobarbituric acid reactive substances (TBARS) - biomarker of lipid peroxidation.
Endocan | Day 1.
  Serum sample collection for ELISA measurement of serum endocan level - proteoglycan associated with endothelium activation

OTHER OUTCOMES:
Blood pressure | Day 1.
  Automatic oscillometric measurement of blood pressure (in mmHg)
Heart rate | Day 1.
  Automatic oscillometric measurement of heart rate (bpm)
Body mass index | Day 1.
  Measurement of body weight (kg) and body height (cm) from which will be combined to report body mass index (BMI) using formula: weight (kg) / [height (m)]2 (kg/m2)
Body composition - Fat Free Mass estimation | Day 1.
  Body composition status measured by a fourterminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically dervide formulas (the original manufacturer's software) will be used to calculate the estimated Fat Free Mass (FFM kg)
Body composition - Fat estimation | Day 1.
  Body composition status measured by a fourterminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically dervide formulas (the original manufacturer's software) will be used to calculate the estimated Fat (Fat Mass kg)
Body fluid status | Day 1.
  Body fluid status measurement by a four-terminal portable impedance analyzer. Based on the value of skin resistance (Ohm) empirically derived formulas (the original manufacturer's software) will be used to calculate the estimated Total Body Water (TBW L), Extracellular Water (ECW L), Intracellular Water (ICW L), Plasma Fluid (PF L) and Interstitial Fluid (IF L).

CONTACTS AND LOCATIONS:
Overall Officials: Martina Kos, MD, Principal Investigator — Osijek University Hospital
Locations (1):
- Osijek University Hospital, Osijek, Croatia